CLINICAL TRIAL: NCT01961505
Title: A Randomized Controlled Study to Determine the Effects and Safety of Topical Compound Tripterygium Wilfordii Hook F in Patients With Active Rheumatoid Arthritis.
Brief Title: Topical Compound Tripterygium Wilfordii Hook F for Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, director, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z111107058811104
Record Dates: First submitted 2013-09-23; First posted 2013-10-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Active Rheumatoid Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Tripterygium group (Experimental): Patients were treated with topical compound tripterygium for 1 hour, twice per day. Area dosages were as followed that each 1st to 5th metacarpophalangeal joints (MCPJs), 1st to 5th proximal interphalangeal joints (PIPJs) and wrist was 3 ml, each elbow and ankle was 5 ml, each knee was 10 ml.
  Interventions: Drug: Topical compound tripterygium
- Topical Placebo group (Placebo Comparator): Patients were treated with topical placebo for 1 hour, twice per day. The dosage was the same as the topical tripterygium group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical compound tripterygium — Topical compound tripterygium was applied for the pain and swollen joints on non-woven fabric for 1 hour, twice per day.
  Arms: Topical Tripterygium group
Drug: Placebo — The topical placebo recipe composes viscous agent which matches by the sucrose, and the usage and dosage were the same as the topical compound tripterygium group.
  Arms: Topical Placebo group

SUMMARY:
Rheumatoid Arthritis (RA) is an autoimmune disease that results in a chronic inflammatory disorder that may affect many synovial joints, and may cause serious disability. It has been confirmed that Tripterygium wilfordii Hook F has effects of anti-inflammatory, immunosuppressive and cartilage protection. This is a prospective randomized controlled study to evaluated the efficacy and safety of external application with compound Tripterygium wilfordii Hook F in treating of patients with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of rheumatoid arthritis, as defined by the American Rheumatism Association 1987 Revised Criteria or European League Against Rheumatism criteria (2009).
* Patients must have moderately to severely active RA,and the DAS-28 score should be from 3.2 to 5.1.
* If taking disease modifying antirheumatic drug (DMARDs)(e.g.Methotrexate), subject must have been on a stable dose for ≥ 3 months prior to randomization.
* If taking non-steroidal anti-inflammatory drugs (NSAIDs), subject must have been on a stable dose for ≥ 4 weeks prior to randomization.
* 16 to 65 years old, having signed the informed consent.

Exclusion Criteria:

* Patients who have skin burst or allergies.
* Patients with sever diseases in Cardiovascular, brain, lung, liver, kidney and hematopoietic system.
* Patients who have been treated by tripterygium, hormones or biological agents.
* Patients who have not been treated by DMARDs before.
* Patients who are unwilling to comply with all study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ACR20 criteria | Week 4
  To meet the criteria, a patient must have 20% or greater improvement in both tender and swollen joints (28 tender and 28 swollen joints were assessed) and 20% or greater improvement in 3 or more of the following: the physician's or patient's assessment of global health status, the patient's assessment of pain on a visual analogue scale, the patient's assessment of function using a modified version of the Health Assessment Questionnaire (HAQ), and the ESR or serum C-reactive protein (CRP) level.

SECONDARY OUTCOMES:
ACR50 criteria | Week 4
  To meet the criteria, a patient must have 50% or greater improvement in both tender and swollen joints (28 tender and 28 swollen joints were assessed) and 50% or greater improvement in 3 or more of the following: the physician's or patient's assessment of global health status, the patient's assessment of pain on a visual analogue scale, the patient's assessment of function using a modified version of the Health Assessment Questionnaire (HAQ), and the ESR or serum C-reactive protein (CRP) level.
28-joint count Disease Activity Score (DAS28) | Baselin and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Quan Jiang, Principal Investigator — Guang'anmen Hospital

IPD SHARING:
Plan to Share IPD: No